CLINICAL TRIAL: NCT05046301
Title: Contrast-Enhanced Mammography (CEM) and CEM-Directed Biopsy for the Evaluation of Extensive Suspicious Mammographic Microcalcifications
Brief Title: Contrast-Enhanced Mammography for the Evaluation of Mammographic Microcalcifications
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0501; NCI-2021-08428 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-08-31; First posted 2021-09-16 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Contrast Media

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Diagnostic (contrast-enhanced mammography): Patients complete a questionnaire and undergo collection of a blood sample. Patients undergo CEM.
  Interventions: Procedure: Biospecimen Collection; Other: Contrast Agent; Procedure: Contrast-Enhanced Mammography; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Correlative studies
  Other Names: Biological Sample Collection
Other: Contrast Agent — Given IV
  Other Names: Contrast; Contrast Drugs; contrast material; Contrast Medium
Procedure: Contrast-Enhanced Mammography — Undergo contrast-enhanced mammography
  Other Names: CEM
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates the added role of contrast-enhanced mammography (CEM), as well as imaging and blood biomarkers, for predicting the presence or absence of high-grade ductal carcinoma in situ (DCIS) or invasive cancer on pathology. Screening mammography is the mainstay of population-wide early breast cancer detection, and mammography-detected cancers are usually of an earlier stage, giving women the best chance of survival. However, the main drawbacks of this type of screening are false positive results and potential over-diagnosis of breast cancer. Suspicious microcalcifications detected with mammography pose a particular diagnostic problem, as they may be associated with invasive and high-grade in-situ cancers like DCIS, but are more often benign or require further workup to verify diagnosis. As such, microcalcifications detected by mammography pose a risk of both over-diagnosis and underestimation of disease severity. This study evaluates the impact of using CEM, compared to standard full field digital mammography (FFDM) for the management of suspicious microcalcifications and prediction of breast cancer in women with this finding.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the added value of contrast enhancement of CEM compared to two dimensional (2D) mammography in predicting invasive malignancy or high-grade DCIS in patients with suspicious mammographic microcalcifications.

SECONDARY OBJECTIVES:

I. To evaluate the added value of contrast enhancement in CEM by comparing the sensitivity/specificity of contrast enhancement to the sensitivity/specificity of FFDM.

II. To evaluate whether the absence of contrast enhancement can predict the absence of high grade DCIS or invasive cancer by establishing the negative predictive value (NPV) of contrast enhancement and comparing it to the NPV of FFDM.

III To evaluate whether the presence of abnormal contrast enhancement can predict the presence of high grade DCIS or invasive malignancy by establishing the positive predictive value (PPV) of contrast enhancement and comparing it to the PPV of FFDM.

IV. To evaluate the influence of the morphology, distribution, and extent of mammographic microcalcifications on the presence and intensity of contrast enhancement.

V. To evaluate the cancer detection rate and the outcomes (need for additional imaging, biopsies, and final pathologic results) of incidental CEM findings.

EXPLORATORY OBJECTIVES:

I. To evaluate the correlation of blood biomarkers and the presence of invasive cancer and high-grade DCIS on pathology in the study patients.

II. To evaluate the technical feasibility of using CEM-guided or CEM-directed stereotactic biopsies in patients with suspicious microcalcifications equal to or exceeding 4 cm in diameter.

III. In patients who undergo CEM targeted or CEM directed biopsy we will evaluate the upgrade rate of DCIS to invasive malignancy or high grade lesions to in-situ or invasive cancer for those patients who will require surgery as a part of their routine clinical care.

IV. To compare the performance of FFDM (obtained as a part of the recent prior screening or diagnostic mammographic work-up) and LE CEM images (obtained as a part of the CEM study) in terms of accuracy, sensitivity, specificity, PPV and NPV.

OUTLINE:

Patients complete a questionnaire and undergo collection of a blood sample. Patients receive contrast intravenously (IV) and undergo CEM.

After completion of study, patients are followed for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Women with suspicious mammographic microcalcifications (Breast Imaging Reporting and Data System [BI-RADS] categories 4 or 5) occupying an area equal to or exceeding 4 cm in diameter and recommended for a stereotactic biopsy, who underwent their diagnostic imaging work-up resulting in a biopsy recommendation at MD Anderson Cancer Center (MDACC) or at an outside facility with a technically acceptable quality of diagnostic mammography, and who are planning to have their stereotactic biopsy at MDACC.
* Age 25-85 years
* Willing to participate in the study, undergo an intravenous (IV) placement, able to undergo iodinated contrast injection, and able to provide informed consent

Exclusion Criteria:

* Reported history of an allergic reaction to iodinated contrast
* History of anaphylactic reaction to any substance that required hospitalization or IV placement in a patient with no known prior uneventful exposure to iodine-based IV contrast
* Renal insufficiency
* Pregnancy or lactation within 6 months
* Breast surgery affecting the site of interest within prior 6 months
* Breast biopsy at the site of interest within the last 2 months
* Mammographic mass or architectural distortion associated with the calcifications in question

Ages: 25 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspicious mammographic microcalcifications
Sampling Method: Non-Probability Sample
Enrollment: 151 (Estimated)
Dates: Start 2021-03-23 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Accuracy | Up to 1 year
  Determined by comparing the contrast-enhanced mammography (CEM)/full field digital mammography (FFDM) results to those of the pathologic evaluations. Specifically, it is defined as the number of concordant cases between CEM/FFDM and pathologic evaluation divided by the total sample size. Descriptive statistics will be used to summarize clinical variables of interest. Specifically, categorical measures will be summarized using frequencies and percentages, and continuous measures will be summarized using means, standard deviations, medians, and ranges.

CONTACTS AND LOCATIONS:
Overall Officials: Olena Weaver, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org